CLINICAL TRIAL: NCT01261533
Title: The Multi-center Exploratory Clinical Trials for the Evaluation of Flexibility, Efficacy, and Safety of a Foldable Capsular Vitreous Body in the Treatment of Severe Retinal Detachment
Brief Title: Flexibility, Efficacy, and Safety of a Foldable Capsular Vitreous Body in the Treatment of Severe Retinal Detachment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GuangZhou WeiShiBo Biotechnology Co., ltd (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISBOR-61165995002
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Retinal Detachment
Keywords: vitreous body substitute; foldable capsular vitreous body
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FCVB team (Experimental): the vitreous cavity is tamponaded with the foldable capsular vitreous body (FCVB)
  Interventions: Device: foldable capsular vitreous body(FCVB)

INTERVENTIONS:
Device: foldable capsular vitreous body(FCVB) — FCVB with silicone oil inside is tamponaded into the vitreous cavity
  Other Names: FCVB

SUMMARY:
The purpose of this study is to determine the feasibility, primary safety and efficacy of foldable capsular vitreous body (FCVB) in the treatment of retinal detachment, based on the multi-center clinical trial.

DETAILED DESCRIPTION:
Previous clinical trial have demonstrated that foldable artificial vitreous body (FCVB),with balanced salt solution (BSS) filled in 11 patients during three-months observation,or silicone oil filled in 4 patients during a six-month observation respectively, can be transplanted into the vitreous body easily, and performances good safety and efficacy in the treatment of severe retinal detachment.

Current multi-center clinical trial was to determine the feasibility, primary safety and efficacy of FCVB with silicone oil filled in the treatment of retinal detachment in 120 patients.

ELIGIBILITY:
Inclusion Criteria:

1. age range from 18 to 65, Refractive error less than ±3D
2. Corrected visual acuity less than 0.05
3. ocular axial length is 16 to 25mm
4. severe retinal detachment that can not be treated by current artificial vitreous body:

   1. Severe unilateral ocular perforating injuries, compounded retinal or choroidal detachments resulted from retinal rupture or retinal choroidal hemorrhage.
   2. Severe unilateral ocular rupture injuries result in retina or choroid defect.
   3. Giant posterior scleral rupture injuries that can not be repaired.
   4. Silicone oil can't be taken out for a long time with incomplete reattachment.
   5. Participants have undergone retinal detachment surgery and silicone oil tamponade twice or more, however, retina is re-detachment after silicone oil removal.
5. Participants can understand the aim of this clinical trial and sign the informed consent form

Exclusion Criteria:

1. Participants have a silica gel allergy or scar diathesis
2. entophthalmia
3. uveitis
4. The contralateral eye suffered from intraocular surgery
5. uncontrollable the other eye diseases
6. Corrected visual acuity of contralateral eye less than 0.4
7. Proliferative diabetic retinopathy
8. the lens of target eye is transparent
9. Serious heart, lung, liver and kidney dysfunction
10. pregnancy, preparation for pregnancy during clinical trial and breast-feeding female
11. drug abuse or alcoholism
12. participated the other drug or medical devices clinical trial before screening of this trial
13. Any research doctors consider that the condition of participants will hinder the clinical trial--Prone to mental stress, loss control of mood, depression etc.
14. Patient adherence is so poor that study procedures can not be finished

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Complete retinal reattach rate at the 52 weeks after implantation of the FCVB | 52 weeks after implantation of the FCVB

SECONDARY OUTCOMES:
Retinal reattach rate, Visual function，and Silicone oil change | Before surgery, 3days,1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks after FCVB implantation surgery (If patients ask for the delay of removal of FCVB, the patients must received a review every three months)
  visual acuity, intraocular pressure, axial length, ocular inflammatory response, the number of corneal endothelial, emulsification rate of silicone oil, migration of silicone oil droplets into the anterior, chamber, anterior chamber angle and ciliary body change, morphological changes of the ocular and FCVB.

CONTACTS AND LOCATIONS:
Overall Officials: Qianying Gao, MD,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - The 2nd affiliated hospital of Harbin Medicinal University., Harbin, Heilongjiang
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Eye and ENT Hospital of FuDan University, Shanghai, Shanghai Municipality
  - XiJing Hospital, Xian, Shanxi
  - The affiliated Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

REFERENCES:
- [Background] Gao Q, Mou S, Ge J, To CH, Hui Y, Liu A, Wang Z, Long C, Tan J. A new strategy to replace the natural vitreous by a novel capsular artificial vitreous body with pressure-control valve. Eye (Lond). 2008 Mar;22(3):461-8. doi: 10.1038/sj.eye.6702875. Epub 2007 May 25. PMID 17525767
- [Background] Gao Q, Chen X, Ge J, Liu Y, Jiang Z, Lin Z, Liu Y. Refractive shifts in four selected artificial vitreous substitutes based on Gullstrand-Emsley and Liou-Brennan schematic eyes. Invest Ophthalmol Vis Sci. 2009 Jul;50(7):3529-34. doi: 10.1167/iovs.08-2802. Epub 2009 Mar 5. PMID 19264881
- [Background] Liu Y, Jiang Z, Gao Q, Ge J, Chen J, Cao X, Shen Q, Ma P. Technical standards of a foldable capsular vitreous body in terms of mechanical, optical, and biocompatible properties. Artif Organs. 2010 Oct;34(10):836-45. doi: 10.1111/j.1525-1594.2010.01006.x. PMID 20618225
- [Background] Liu Y, Ke Q, Chen J, Wang Z, Xie Z, Jiang Z, Ge J, Gao Q. Sustained mechanical release of dexamethasone sodium phosphate from a foldable capsular vitreous body. Invest Ophthalmol Vis Sci. 2010 Mar;51(3):1636-42. doi: 10.1167/iovs.09-4134. Epub 2009 Oct 15. PMID 19834025
- [Background] Lin X, Ge J, Gao Q, Wang Z, Long C, He L, Liu Y, Jiang Z. Evaluation of the flexibility, efficacy, and safety of a foldable capsular vitreous body in the treatment of severe retinal detachment. Invest Ophthalmol Vis Sci. 2011 Jan 21;52(1):374-81. doi: 10.1167/iovs.10-5869. PMID 20811065
- [Background] Zhang R, Wang T, Xie C, Lin X, Jiang Z, Wang Z, Liu Y, Luo Y, Long C, He L, Wang P, Gao Q. Evaluation of supporting role of a foldable capsular vitreous body with magnetic resonance imaging in the treatment of severe retinal detachment in human eyes. Eye (Lond). 2011 Jun;25(6):794-802. doi: 10.1038/eye.2011.61. Epub 2011 Mar 18. PMID 21423138
- [Background] Wang P, Gao Q, Jiang Z, Lin J, Liu Y, Chen J, Zhou L, Li H, Yang Q, Wang T. Biocompatibility and retinal support of a foldable capsular vitreous body injected with saline or silicone oil implanted in rabbit eyes. Clin Exp Ophthalmol. 2012 Jan-Feb;40(1):e67-75. doi: 10.1111/j.1442-9071.2011.02664.x. Epub 2011 Oct 20. PMID 21883770
- [Background] Lin X, Wang Z, Jiang Z, Long C, Liu Y, Wang P, Jin C, Yi C, Gao Q. Preliminary efficacy and safety of a silicone oil-filled foldable capsular vitreous body in the treatment of severe retinal detachment. Retina. 2012 Apr;32(4):729-41. doi: 10.1097/IAE.0b013e31822b1f80. PMID 22105508